CLINICAL TRIAL: NCT01686451
Title: Comparison Between XueZhiKang and Simvastatin on Fatigue: a Single-center, Randomized Clinical Trial
Brief Title: The Effect of XueZhiKang on Fatigue：Comparing With Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, JiFei Tang, Director, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Wenzhou
Record Dates: First submitted 2012-09-03; First posted 2012-09-18 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — xuezhikang; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XueZhiKang (Experimental): Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
  Interventions: Drug: XueZhiKang
- Simvastatin (Active Comparator): Participants will receive 20mg of simvastatin daily for 4 weeks.
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: XueZhiKang — Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
  Arms: XueZhiKang
Drug: simvastatin — Participants will receive 20mg of simvastatin daily for 4 weeks.
  Other Names: shujiangzhi
  Arms: Simvastatin

SUMMARY:
Both XueZhiKang and Statins are cholesterol-lowering medications that are often prescribed for individuals with high cholesterol and who are at risk for cardiovascular disease (CVD). Several studies, including one randomized, double-blind, placebo-controlled clinical trial, have suggested that the use of statins is more frequently associated with fatigue. And XueZhiKang may be not. The purpose of this study is to compare the effect of these two medications on fatigue in persons who are at moderate to low CVD risk based on the risk estimation system in ESC(European Society of Cardiology)/ESA(European Atherosclerosis Society) guidelines (2011) for the management of dyslipidemias.

DETAILED DESCRIPTION:
Individuals at risk for cardiovascular disease (CVD) are often prescribed statins, which are medications that reduce the amount of cholesterol in the blood. By lowering cholesterol levels, these individuals have a lower incidence of coronary artery disease, ischemic stroke, and peripheral arterial disease and so on. While statins are effective at lowering cholesterol levels, their effect on fatigue is obvious and has been suggested by several studies, including one randomized, double-blind, placebo-controlled clinical trial. And XueZhiKang may be not. The purpose of this study is to compare the effect of these two medications on fatigue in persons who are at moderate to low CVD risk based on the risk estimation system in ESC(European Society of Cardiology)/ESA(European Atherosclerosis Society) guidelines (2011) for the management of dyslipidemias.

This study will enroll individuals who do not currently take cholesterol-lowering medications. Participants will be randomly assigned to receive 600mg of XueZhiKang twice a day, or 20mg of simvastatin daily for 4 weeks. Study visits will occur at baseline and Week 4. Blood will be collected for laboratory testing, and standardized psychological questionnaires will assess fatigue scores and physical activity levels at baseline and week 4. Pill count will be used to assess adherence of XueZhiKang and simvastatin treatment at week 4. At week 4, medication side effects will be monitored and tests of alanine aminotransferase (ALT), aspartate aminotransaminase (AST) and creatine phosphate kinase (CPK) will be performed. At week 4, medication efficacy will be assessed and test of low-density lipoprotein cholesterol (LDL-C) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. LDL cholesterol level between 115-190 mg/dL;
2. Able to fast prior to blood draw;
3. Able to comfortably read and write in Chinese;
4. Able and willing to refrain from donating whole blood during study participation;
5. Willing to abstain from consuming large amounts of grapefruit juice.

Exclusion Criteria:

1. Current use of lipid-lowering medications;
2. Documented cardiovascular disease (CVD) by invasive or non-invasive testing (such as coronary angiography, nuclear imaging, stress echocardiography, carotid plaque on ultrasound), previous myocardial infarction (MI), acute coronary syndrome (ACS), coronary revascularization [percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)] and other arterial revascularization procedures, ischaemic stroke, peripheral arterial disease(PAD);
3. Patients with type 2 diabetes, patients with type 1 diabetes with target organ damage (such as microalbuminuria);
4. Patients with moderate to severe chronic kidney disease [glomerular filtration rate (GFR) < 60 mL/min/1.73㎡];
5. Markedly elevated single risk factors such as familial dyslipidaemias and severe hypertension;
6. A calculated SCORE ≥5% for 10 year risk of fatal CVD;
7. Cancer;
8. HIV infected;
9. Medical or psychiatric condition that prevents full study participation or follow-up (e.g., active psychosis);
10. Active liver disease or unexplained persistent elevated transaminase levels；
11. Major surgery or hospitalization in the 3 months prior to study entry;
12. Current use of cyclosporin, erythromycin, clarithromycin, nefazodone, or any "azole" antifungals, including fluconazole, itraconazole, ketoconazole, mibefradil, or protease inhibitors;
13. Female of childbearing potential;
14. Current participation in another clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jifei Tang, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Second Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Xue Y, Tao L, Wu S, Wang G, Qian L, Li J, Liao L, Tang J, Ji K. Red yeast rice induces less muscle fatigue symptom than simvastatin in dyslipidemic patients: a single center randomized pilot trial. BMC Cardiovasc Disord. 2017 May 18;17(1):127. doi: 10.1186/s12872-017-0560-z. PMID 28521773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 10, 2012, through September 15, 2013, 243 patients were screened and 60 patients who met the inclusion criteria were enrolled and randomly assigned to either simvastatin (33 patients) or xuezhikang (27 patients) at medical clinic.
Pre-assignment Details: 183 eligible patients were excluded with 160 patients declined to participate while 19 patients were currently using lipid-lowering medications, 3 patients were suffering from chronic kidney disease or active liver disease and 1 was of currently childbearing.
Groups:
- Simvastatin: Participants will receive 20mg of simvastatin daily for 4 weeks.
  simvastatin : Participants will receive 20mg of simvastatin daily for 4 weeks.
- XueZhiKang: Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
  XueZhiKang : Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
Period: Overall Study
Arm/Group | Simvastatin | XueZhiKang
Started | 33 | 27
Completed | 33 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 60 patients with dyslipidemia and moderate to low cardiovascular disease (CVD) risk were randomly assigned in an open label fashion to receive either simvastatin (n=33) 20 mg daily or xuezhikang (n=27) 600 mg twice daily. All 60 patients were included in baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | XueZhiKang | Total
Number analyzed (Participants) | 33 | 27 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 27 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.18 (7.00) | 47.04 (5.83) | 46.57 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  China | 33 | 27 | 60
Current cigarette smoker, Categorical [Number; unit: participants]
  Current cigarette smoker | 3 | 2 | 5
  Not Current cigarette smoker | 30 | 25 | 55
Arterial hypertension, Categorical [Number; unit: participants]
  Arterial hypertension | 26 | 16 | 42
  Not Arterial hypertension | 7 | 11 | 18
Arterial blood pressure, Continuous [Mean (Standard Deviation); unit: mmHg]
  Systolic blood pressure | 148.06 (18.51) | 147.89 (17.03) | 147.98 (17.71)
  Diastolic blood pressure | 84.18 (6.95) | 83.00 (8.82) | 83.65 (7.80)
Fasting blood glucose, Continuous [Mean (Standard Deviation); unit: mmol/L] | 5.10 (0.36) | 5.33 (0.52) | 5.20 (0.45)
Triglyceride, Continuous [Mean (Standard Deviation); unit: mmol/L] | 1.76 (1.00) | 1.61 (0.65) | 1.69 (0.86)
Total cholesterol, Continuous [Mean (Standard Deviation); unit: mmol/L] | 5.91 (0.71) | 5.82 (0.73) | 5.87 (0.72)
High-density lipoprotein-cholesterol, Continuous [Mean (Standard Deviation); unit: mmol/L] | 1.27 (0.25) | 1.23 (0.25) | 1.26 (0.25)
Low-density lipoprotein-cholesterol, Continuous [Mean (Standard Deviation); unit: mmol/L] | 3.72 (0.48) | 3.74 (0.55) | 3.73 (0.50)
Alanine aminotransferase, Continuous [Mean (Standard Deviation); unit: U/L] | 28.58 (10.55) | 30.33 (13.30) | 29.37 (11.79)
Aspartate aminotransferase, Continuous [Mean (Standard Deviation); unit: U/L] | 24.12 (7.00) | 25.63 (7.53) | 24.80 (7.22)
Creatine phosphate kinase, Continuous [Mean (Standard Deviation); unit: U/L] | 80.82 (24.91) | 91.65 (23.71) | 85.69 (24.78)
Creatinine, Continuous [Mean (Standard Deviation); unit: μmol/L] | 72.57 (14.44) | 75.59 (17.20) | 73.93 (15.68)
Fatigue score, Continuous [Mean (Standard Deviation); unit: units on a scale] — The fatigue score was assessed by a fatigue questionnaire named as Fatigue Assessment Scale (FAS) which used 10-item fatigue measure with the fatigue score ranged from 10-50. The higher score was meaning of higher level of fatigue.
  units on a scale | 19.58 (2.55) | 19.26 (1.85) | 19.43 (2.25)
Physical activity level, Categorical [Number; unit: participants] — We estimated physical activity level by short version of international physical activity questionnaire (IPAQ) with categorical score ranged from low to high. The higher score was meaning of lower physical activity level.
  participants
    Low level | 14 | 3 | 17
    Moderate level | 10 | 12 | 22
    High level | 9 | 12 | 21

OUTCOME MEASURES:

1. Secondary Outcome: Treatment Efficacy
Description: Treatment efficacy was estimated on the basis of triglyceride (TG), total cholesterol (TC), high-density lipoprotein-cholesterol (HDL-C), as well as LDL-C levels obtained at baseline and week 4.
Time Frame: Measured at baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Simvastatin/Baseline; Simvastatin/Week 4: Participants will receive 20mg of simvastatin daily for 4 weeks.
  simvastatin : Participants will receive 20mg of simvastatin daily for 4 weeks.
- XueZhiKang/Baseline; XueZhiKang/Week 4: Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
  XueZhiKang : Participants will receive 600mg of XueZhiKang twice a day for 4 weeks.
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
mmol/L
  TG level at baseline and week 4 | 1.76 (1.00) | 1.54 (1.01) | 1.61 (0.65) | 1.36 (0.69)
  TC level at baseline and week 4 | 5.91 (0.71) | 4.73 (1.08) | 5.82 (0.73) | 4.72 (1.16)
  HDL level at baseline and week 4 | 1.27 (0.25) | 1.32 (0.36) | 1.23 (0.25) | 1.37 (0.44)
  LDL level at baseline and week 4 | 3.72 (0.48) | 2.54 (0.72) | 3.74 (0.55) | 2.45 (0.71)

2. Primary Outcome: Comparison Between XueZhiKang and Simvastatin on Fatigue Scores
Description: At baseline and week 4, the fatigue score was assessed by a fatigue questionnaire named as Fatigue Assessment Scale (FAS) which used 10-item fatigue measure with the fatigue score ranged from 10-50. The higher score was meaning of higher level of fatigue.
Time Frame: Measured at baseline and week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
units on a scale | 19.58 (2.55) | 21.58 (2.75) | 19.26 (1.85) | 19.33 (1.90)

3. Other Pre Specified Outcome: Comparison of XueZhiKang With Simvastatin of Physical Activity Level
Description: At baseline and week 4, we estimated physical activity level by short version of international physical activity questionnaire (IPAQ) with categorical score ranged from low to high. The higher score was meaning of lower physical activity level.
Time Frame: Measured at baseline and week 4
Measure: Number; unit: participants
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
participants
  Low level at baseline and week 4 | 14 | 25 | 3 | 3
  Moderate level at baseline and week 4 | 10 | 8 | 12 | 15
  High level at baseline and week 4 | 9 | 0 | 12 | 9

4. Other Pre Specified Outcome: Comparison of Safety Laboratory Testings (ALT,AST,CPK) Between Simvastatin- and Xuezhikang-groups
Description: Fasting blood samples were collected at weeks 0 (randomization) and 4 (end of study) for clinical chemistry.
Time Frame: Measured at baseline and week 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
U/L
  ALT level at baseline and week 4 | 28.58 (10.55) | 28.73 (13.10) | 30.33 (13.30) | 28.67 (14.73)
  AST level at baseline and week 4 | 24.12 (6.99) | 24.42 (6.89) | 25.63 (7.53) | 25.85 (7.24)
  CPK level at baseline and week 4 | 80.82 (24.91) | 82.76 (33.80) | 91.65 (23.71) | 90.92 (24.36)

5. Other Pre Specified Outcome: Comparison of Safety Laboratory Testing (Cr) Between Simvastatin- and Xuezhikang-group
Description: Fasting blood samples were collected at weeks 0 (randomization) and 4 (end of study) for clinical chemistry.
Time Frame: Measured at baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
mmol/L | 72.57 (14.44) | 71.95 (14.34) | 75.59 (17.20) | 76.51 (16.39)

6. Other Pre Specified Outcome: Treatment Adherence at Week 4 in Simvastatin- and Xuezhikang-group
Description: We counted the total number of pills that were dispensed to the participants at baseline and the total number of pills that were taken by participants at week 4.
Time Frame: Measured at baseline and week 4
Measure: Number; unit: number of pills
Arm/Group | Simvastatin/Baseline | Simvastatin/Week 4 | XueZhiKang/Baseline | XueZhiKang/Week 4
Number analyzed (Participants) | 33 | 33 | 27 | 27
number of pills | 462 | 462 | 3024 | 3024

ADVERSE EVENTS:
Arm/Group | Simvastatin | XueZhiKang
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/27
Other Adverse Events (participants affected / at risk) | 0/33 | 0/27

LIMITATIONS AND CAVEATS:
There are some limitations to this research. First, the sample size was relative small. Second, the follow-up period was short (4 weeks).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less